CLINICAL TRIAL: NCT07109076
Title: Effect of Immediate Skin-to-Skin Contact With the Mother on Heart Rate Variability in Newborns After Cesarean Secton
Brief Title: Effect of Immediate Skin-to-Skin Contact on Neonatal Heart Rate Variability After Cesarean Secton
Acronym: HRV-SCENE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miha Lucovnik, Professor Miha Lucovnik, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0120-227/2025-2711-4
Record Dates: First submitted 2025-07-03; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Adaptation
Keywords: heart rate variability; cesarean section; cesarean birth; skin-to-skin contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skin-to-skin contact group (Experimental): Uninterrupted skin-to-skin contact between the neonate and the mother will be initiated immediately and maintained for at least 15 minutes following cesarean birth.
  Interventions: Other: skin-to-skin contact
- control group (Active Comparator): Neonates and mother in this arm will receive routine postnatal care without early skin-to-skin contact. Current routine neonatal care following cesarean section includes delayed umbilical cord clamping. Afterward, the newborn is dried by a midwife, dressed, briefly shown to the mother, and then handed over to the father.
  Interventions: Other: routine care

INTERVENTIONS:
Other: skin-to-skin contact — Uninterrupted skin-to-skin contact between the neonate and the mother will be initiated immediately and maintained for at least 15 minutes following cesarean birth.
  Arms: skin-to-skin contact group
Other: routine care — Current routine neonatal care following cesarean section includes delayed umbilical cord clamping. Afterward, the newborn is dried by a midwife, dressed, briefly shown to the mother, and then handed over to the father.
  Arms: control group

SUMMARY:
At birth, both the newborn and the mother experience adaptive stress, which can be measured using objective physiological methods. One of the possible methods is monitoring heart rate variability, which is an indirect indicator of the balance between the sympathetic and parasympathetic branches of the autonomic nervous system. The proposed study will monitor the effect of early skin-to-skin contact on heart rate variability in newborns delivered by cesarean section and their mothers.

The researchers hypothesize that newborns and mothers who are provided with immediate direct skin-to-skin contact, compared to the control group receiving standard care, will exhibit higher heart beat-to-beat interval variability in the first hours after birth. This is expected to result from reduced stress and activation of the parasympathetic nervous system.

The study will include 80 newborn-mother pairs with a gestational age of 39 weeks or more, delivered via planned cesarean section. Participants will be randomly assigned to a study group (skin-to-skin contact lasting at least 15 minutes after cesarean birth) and a control group (standard care), with 40 newborns in each group. Maternal and neonatal ECG will be monitored for 15 minutes following cesarean birth in both groups. In addition, neonatal ECG will be monitored at 6, 12 and 24 hours postpartum. Time-domain analyses of hearth rate variability will be performed.

DETAILED DESCRIPTION:
At the time of birth, both the newborn and the mother undergo a complex and dynamic process of physiological and psychological adaptation, often referred to as perinatal adaptive stress. This adaptive stress response involves significant alterations in neuroendocrine and autonomic function, including activation of the hypothalamic-pituitary-adrenal (HPA) axis and fluctuations in autonomic nervous system (ANS) activity. These physiological responses can be objectively assessed using various biomarkers and physiological parameters. Among the most informative and non-invasive indicators of autonomic regulation is heart rate variability (HRV)-a measure of the variation in time intervals between consecutive heartbeats (RR intervals), which reflects the interplay between the sympathetic and parasympathetic branches of the ANS.

HRV has been widely used in neonatal and maternal research as a surrogate marker of stress, resilience, and autonomic function. High HRV is generally associated with enhanced parasympathetic (vagal) tone and a more flexible and adaptive physiological state, whereas low HRV is indicative of stress, reduced vagal activity, and sympathetic predominance. The immediate postpartum period, particularly following cesarean delivery, represents a critical window during which both maternal and neonatal physiological systems transition from intrauterine to extrauterine life, often in the absence of the hormonal and mechanical stimuli associated with vaginal delivery.

The proposed randomized controlled trial aims to investigate the effect of early skin-to-skin contact (SSC) between mother and newborn on HRV in both participants following planned cesarean section. Early SSC has been shown in previous studies to promote maternal-infant bonding, thermoregulation, breastfeeding initiation, and physiological stability; however, its impact on autonomic modulation as assessed by HRV-particularly in cesarean births-remains underexplored.

The central hypothesis of this study is that immediate and sustained skin-to-skin contact will result in significantly greater HRV in both neonates and mothers, as compared to a control group receiving standard post-cesarean care. This increase in HRV is expected to reflect reduced perinatal stress, enhanced vagal activation, and improved autonomic balance during the early postpartum period.

The study will enroll 80 mother-newborn dyads with a gestational age of ≥39 weeks undergoing elective cesarean section. Participants will be randomly assigned to either the intervention group, in which uninterrupted skin-to-skin contact will be initiated immediately and maintained for at least 15 minutes following birth, or the control group, which will receive routine postnatal care without early SSC. Each group will comprise 40 dyads.

Electrocardiographic (ECG) monitoring will be conducted in both mothers and newborns during the first 15 minutes following birth to capture real-time cardiac data. In addition, neonatal ECG will be monitored at 6, 12 and 24 hours postpartum. HRV will be analyzed using time-domain methods, in accordance with established international standards.

ELIGIBILITY:
Inclusion Criteria:

* planned cesarean section
* gestational age 39 weeks 0/7 or more

Exclusion Criteria:

* Pregnancy complications (e.g. hypertensive disorders in pregnancy, fetal growth restriction, etc.)
* neonatal resuscitation at birth

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Neonatal RMSSD 15 minutes after birth | 15 minutes following cesarean birth.
  RMSSD is a time-domain HRV measure. It is defined as the square root of the mean of the squares of successive differences between adjacent normal (NN) heartbeats (i.e., RR intervals) and expressed in milliseconds (ms).
Neonatal SDNN 15 minutes after birth | 15 minutes following cesarean birth
  SDNN is a time-domain HRV measure. It is defined as the standard deviation of all normal-to-normal (NN) RR intervals over the recorded period and expressed in milliseconds (ms).
Neonatal pNN50 15 minutes after birth | 15 minutes following cesarean birth
  pNN50 is a time-domain HRV measure. It is defined as the percentage of successive NN (normal-to-normal) intervals that differ from each other by more than 50 milliseconds.

SECONDARY OUTCOMES:
Maternal RMSSD 15 minutes after birth | 15 minutes following cesarean birth
  RMSSD is a time-domain HRV measure. It is defined as the square root of the mean of the squares of successive differences between adjacent normal (NN) heartbeats (i.e., RR intervals) and expressed in milliseconds (ms).
Maternal SDNN 15 minutes after birth | 15 minutes following cesarean birth
  SDNN is a time-domain HRV measure. It is defined as the standard deviation of all normal-to-normal (NN) RR intervals over the recorded period and expressed in milliseconds (ms).
Maternal pNN50 15 minutes after birth | 15 minutes following cesarean birth
  pNN50 is a time-domain HRV measure. It is defined as the percentage of successive NN (normal-to-normal) intervals that differ from each other by more than 50 milliseconds.
Neonatal RMSSD 6 hours after birth | 6 hours after cesarean birth
  RMSSD is a time-domain HRV measure. It is defined as the square root of the mean of the squares of successive differences between adjacent normal (NN) heartbeats (i.e., RR intervals) and expressed in milliseconds (ms).
Neonatal SDNN 6 hours after birth | 6 hours after cesarean birth
  SDNN is a time-domain HRV measure. It is defined as the standard deviation of all normal-to-normal (NN) RR intervals over the recorded period and expressed in milliseconds (ms).
Neonatal pNN50 6 hours after birth | 6 hours after cesarean birth
  pNN50 is a time-domain HRV measure. It is defined as the percentage of successive NN (normal-to-normal) intervals that differ from each other by more than 50 milliseconds.
Neonatal RMSSD 12 hours after birth | 12 hours after cesarean birth
  RMSSD is a time-domain HRV measure. It is defined as the square root of the mean of the squares of successive differences between adjacent normal (NN) heartbeats (i.e., RR intervals) and expressed in milliseconds (ms).
Neonatal SDNN 12 hours after birth | 12 hours after cesarean birth
  SDNN is a time-domain HRV measure. It is defined as the standard deviation of all normal-to-normal (NN) RR intervals over the recorded period and expressed in milliseconds (ms).
Neonatal pNN50 12 hours after birth | 12 hours after cesarean birth
  pNN50 is a time-domain HRV measure. It is defined as the percentage of successive NN (normal-to-normal) intervals that differ from each other by more than 50 milliseconds.
Neonatal RMSSD 24 hours after birth | 24 hours after cesarean birth
  RMSSD is a time-domain HRV measure. It is defined as the square root of the mean of the squares of successive differences between adjacent normal (NN) heartbeats (i.e., RR intervals) and expressed in milliseconds (ms).
Neonatal SDNN 24 hours after birth | 24 hours after cesarean birth
  SDNN is a time-domain HRV measure. It is defined as the standard deviation of all normal-to-normal (NN) RR intervals over the recorded period and expressed in milliseconds (ms).
Neonatal pNN50 24 hours after birth | 24 hours after cesarean birth
  pNN50 is a time-domain HRV measure. It is defined as the percentage of successive NN (normal-to-normal) intervals that differ from each other by more than 50 milliseconds.

OTHER OUTCOMES:
Neonatal-maternal hearth rate phase synchronisation | 15 minutes after cesarean birth
  Phase synchronisation between neonatal and maternal heart rate in the first 15 minutes after birth will be expressed as a phase synchronisation index (values between 0 (no synchronisation) and 1 (perfect synchronisation)).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be stored and shared upon request.